CLINICAL TRIAL: NCT04570917
Title: Effectiveness of an Online Educational Intervention to Reduce Ageism in Undergraduate Students in an Entry-level Nutrition Class
Brief Title: Online Education Intervention to Reduce Ageism Among Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi, Oxford (Other)
Responsible Party: Principal Investigator, Nadeeja Wijayatunga, Assistant Professor, University of Mississippi, Oxford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21x-046
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-11

CONDITIONS: Ageism
Keywords: Ageism; Older adults; Educational intervention
MeSH Terms: conditions — Ageism

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (INT) (Experimental): An online learning module targeted to reduce ageism will be delivered to the INT group.
  Interventions: Behavioral: Online educational intervention to reduce ageism
- Control group (CON) (Active Comparator): An online learning module on diversity and cultural competence will be delivered to the CON group.
  Interventions: Behavioral: Online educational intervention to enhance cultural competance

INTERVENTIONS:
Behavioral: Online educational intervention to reduce ageism — Participants in this group will go over multiple short videos covering the following content:1). Myths about aging, 2). Ageism and its negative effects, 3). Distorted views about aging among young adults, 4). Ageism during the COVID-19 pandemic, and 5). importance of reducing ageism among healthcare professionals. These will be multiple videos posted on the LMS (Blackboard). At the end of the lesson, they will be asked to briefly write what they learned on Blackboard as an assignment.
  Arms: Intervention group (INT)
Behavioral: Online educational intervention to enhance cultural competance — Participants in the control group will go over multiple short videos covering the following content: 1). Myths about cultural competence, 2) Cultural competence for health care professionals including dietitians, 3). Connecting culture and food, and 4). Importance of cultural competence in sports dietitians. At the end of the lesson, they will be asked to briefly write what they learned. These will be multiple videos posted on the LMS (Blackboard). At the end of the lesson, they will be asked to briefly write what they learned on Blackboard as an assignment.
  Arms: Control group (CON)

SUMMARY:
Ageism is common is healthcare workers, and that results in negative outcomes for elderly patients. This randomized controlled trial is to determine if age bias could be changed by an online learning activity in undergraduate students in an entry-level nutrition class.

DETAILED DESCRIPTION:
This randomized controlled trial with two parallel arms is to determine the effect of an online educational intervention developed to reduce ageism in undergraduate students enrolled in an entry-level Nutrition class. Eligible study participants will be randomized into either the "Intervention group" (INT) or the "Control group" (CON). The two groups will have different learning material delivered online via Blackboard (Learning Management System/LMS). These include a collection of short videos developed by the researchers, as well as relevant videos available on the web. Participants in the INT group will learn about aging and ageism, while the CON group will learn about diversity and cultural competence. Sociodemographic data, percieved risk of COVID-19, preventative behaviors related ot COVID-19 will be collected using a questionnaire at baseline. Ageism will be assessed using standard questionnaires. Data collection will be done at three time points: Pre-intervention, immediate post intervention and 2-weeks post-intervention. Difference between groups for pre-post intervention changes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Enrolled in 3 sections of the introductory level nutrition course taught by three different instructors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Difference between groups for pre-and post intervention changes in the score of Fraboni's Scale for Ageism | From Pre- to immediate post- intervention
  Higher Fraboni's score indicates more bias.
Difference between groups for pre- and 2-weeks post intervention changes in the score of Fraboni's Scale for Ageism | From Pre- to 2-weeks post-intervention
  Higher Fraboni's score indicates more bias.
Difference between groups for pre-post intervention changes in benevolent subscores of the Ambivalent ageism scale | From Pre- to immediate post- intervention
  Higher benevolent score indicates more benevolent ageism
Difference between groups for pre and 2-weeks post intervention changes in benevolent subscores of the Ambivalent ageism scale Higher score indicates more benevolent bias. | From Pre- to 2-weeks post-intervention
  Higher benevolent score indicates more benevolent ageism
Difference between groups for pre-post intervention changes in hostile subscores of the Ambivalent ageism scale | From Pre- to immediate post- intervention
  Higher hostile score indicates more hostile ageism
Difference between groups for pre and 2-week post intervention changes in hostile subscores of the Ambivalent ageism scale | From Pre- to 2-weeks post-intervention
  Higher hostile score indicates more hostile ageism

SECONDARY OUTCOMES:
Difference between groups for pre-post intervention changes in age-related implicit bias | From Pre- to immediate post- intervention
Difference between groups for pre and 2-week post intervention changes in age-related implicit bias | From Pre- to 2-weeks post-intervention
Difference between groups for pre-post intervention changes in the value (years) used to define "old age" | From Pre- to immediate post- intervention
Difference between groups for pre and 2-weeks post intervention changes in the value (years) used to define "old age" | From Pre- to 2-weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nadeeja Wijayatunga, PhD, Principal Investigator — Assistant Professor, Department of Nutrition and Hospitality Management
Locations (1):
- University of Mississippi, Oxford, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the de-identified data on ICPSR database
Time Frame: Within 6 months time after the publication of the primary and secondary analysis planned.
Access Criteria: Public access database
URL: https://www.icpsr.umich.edu/web/pages/index.html